CLINICAL TRIAL: NCT00339222
Title: Family Study of Melanoma in Italy
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902038; 02-C-N038; NCT00556829 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Melanoma; Dysplastic Nevi; Melanocytic Nevi
Keywords: Genetics; Kindreds; Mediterranean Population; Nevi; Pigmentation; Melanoma-Prone Families; Sun Exposure; Melanoma
MeSH Terms: conditions — Melanoma; Dysplastic Nevus Syndrome; Nevus, Pigmented; Nevus

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood, lymphocytes, tissue sections, plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Melanoma-prone families from dermatology clinics.

SUMMARY:
During the course of a case-control study of melanoma conducted at the Bufalini Hospital, Cesena, Italy in the years 1994-1996, 20 families with 2 or 3 melanoma cases were identified and studied. The area where the study was conducted showed the steepest increase in melanoma incidence in Mediterranean populations between the years 1987 and 1997.

Clinical characteristics of melanoma in the families studied were similar to those typically described in fair-skinned populations, but no relevant mutations in the coding regions of known candidate genes from melanoma have been found. Lack of findings could be due to the modest number of families and the small number of affected CMM cases examined. We cannot exclude the possibility of alterations in introns, splicing sites or promoter regions. Also epigenetic factors could affect the expression of the gene products we studied. Alternatively, germline alterations of a gene(s) other than the candidate genes we analyzed may play an important role in melanoma predisposition in this population. A large number of families is needed to test these hypotheses.

These additional families could provide an important contribution to the understanding o melanoma development. In fact, this population does not generally have the host characteristics that are usually associated with higher risk for melanoma (e.g., light skin color, red hair, blue eyes, multiple freckles, tendency to sunburn, etc.) but do have a relative high frequency of dysplastic nevi and melanoma.

The main objective of this study is to recruit more families at the Bufalini Hospital, Cesena, Italy in order to reach a larger sample size. Recently, 16 potential melanoma-prone families have been identified through patient's or physicians' referrals by the Dermatologists at the Bufalini Hospital. The dermatologists have maintained close relationships with members of these families and are confident that these subjects would be willing to participate in a study if contacted. The first goal of our study is to contact this family group and verify their willingness to participate in the study. In addition, new families could be identified and recruited.

We propose to conduct a pilot project. We estimate recruitment of approximately 25 families with 2 or more melanoma cases in first -degree relatives over a one-year period, including the 16 families already identified and approximately 10 new kindreds. At the end of the pilot phase we will determine the feasibility of continuing recruitment.

DETAILED DESCRIPTION:
To date 557 subjects, including cases of melanoma and unaffected relatives, have been recruited in the family study of melanoma at the Bufalini Hospital, Cesena, Italy, University ofl'Aquila, L'Aquila, Italy, and the Istituto Valenciano de Oncologia, Valencia, Spain. Clinical characteristics of melanoma in the families studied were similar to those typically described in fair-skinned populations.

In the original study from the Bufalini Hospital, only 7% of the families analyzed have been shown to carry mutation in the CDKN2A gene, known candidate gene for melanoma, and no other mutation in additional susceptibility genes have been identified. The possibility of alterations in introns, splicing sites, or promoter regions cannot be excluded. Also, epigenetic factors could affect the expression of the gene products we studied. Alternatively, germline alterations of a gene(s) other than the candidate genes may play an important role in melanoma predisposition in this population. We began genome-wide scanning of the first 47 families. There was no evidence for linkage to either chromosome 9 or chromosome 1, previously shown to be susceptibility loci for melanoma. We extended the samples size also including melanoma-prone families from other Italian investigators. We have performed fine mapping of the loci that appeared interesting in the first linkage analysis. We did not confirm the previous association with the disease and published a manuscript to report the null results. Some of these families were also analyzed together with other families worldwide in linkage and genome-wide association studies with the goal of identifying loci potentially important for melanoma etiology. Moreover, some individuals from this study are being analyzed for presence of variants in susceptibility genes in pigmentation, DNA repair, and other pathways together with the melanoma samples from the case-control study (02-C- N(35). Finally, some families with three or more affected individuals are ongoing exomic sequencing with the goal of identifying novel loci associated with melanoma susceptibility. More than 100 subjects have been sequenced to date. We have identified a potentially important candidate gene for melanoma and are investigating additional families and melanoma cases to verify whether we can replicate this finding.

This protocol proposes to continue recruitment of families in order to reach a larger sample size for future analysis. The additional families could provide an important contribution to the understanding of melanoma development.

In addition, this protocol proposes to continue recruiting subjects for the tissue study subgroup at the Bufalini Hospital of Cesena, the Unviersity of I' Aquila, Italy and the Istituto Valenciano de Oncologia, Valencia, Spain. To date, 98 subjects have been enrolled in this study. The study aims at investigating the progression from nevi to melanoma in a cross sectional study of melanoma cases. The tissue study component focuses on the comparison of gene expression, somatic mutations, genetic variants, and proteomics profile in normal skin, common melanocytic nevi, dysplastic nevi, and melanoma tissue samples from the same individuals (familial or sporadic cases). Each subject completes an interview based questionnaire on sun exposure, pigmentation, sunsensitivity, family and medical history, and other melanoma risk factors and donates a blood sample.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals with the diagnosis of CMM at the Department of Dermatology, Bufalini Hospital, Cesena, Italy who have other family members affected with CMM will be eligible for participation.

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Melanoma-prone families from dermatology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1708 (Actual)
Dates: Start 2001-11-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Defining the clinical spectrum and natural history of familial melanoma and susceptibility states over multiple generations | Ongoing
  Melanoma Risk

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Landi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (7):
- Italy (5):
  - Ospedale Maurizio Bufalini Cesena, Italy, Cessana
  - University of Genoa, Genoa
  - University of L'Aquila, L’Aquila
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Oncologico Veneto IRCCS University of Padua, Padua
- Spain (2):
  - Hospital Clinic of Barcelona (Centre de Diagnostic Biomedic), Barcelona
  - Instituto Valenciano de Oncologia, Valencia

REFERENCES:
- [Background] Shi J, Yang XR, Ballew B, Rotunno M, Calista D, Fargnoli MC, Ghiorzo P, Bressac-de Paillerets B, Nagore E, Avril MF, Caporaso NE, McMaster ML, Cullen M, Wang Z, Zhang X; NCI DCEG Cancer Sequencing Working Group; NCI DCEG Cancer Genomics Research Laboratory; French Familial Melanoma Study Group; Bruno W, Pastorino L, Queirolo P, Banuls-Roca J, Garcia-Casado Z, Vaysse A, Mohamdi H, Riazalhosseini Y, Foglio M, Jouenne F, Hua X, Hyland PL, Yin J, Vallabhaneni H, Chai W, Minghetti P, Pellegrini C, Ravichandran S, Eggermont A, Lathrop M, Peris K, Scarra GB, Landi G, Savage SA, Sampson JN, He J, Yeager M, Goldin LR, Demenais F, Chanock SJ, Tucker MA, Goldstein AM, Liu Y, Landi MT. Rare missense variants in POT1 predispose to familial cutaneous malignant melanoma. Nat Genet. 2014 May;46(5):482-6. doi: 10.1038/ng.2941. Epub 2014 Mar 30. PMID 24686846
- [Background] Iles MM, Law MH, Stacey SN, Han J, Fang S, Pfeiffer R, Harland M, Macgregor S, Taylor JC, Aben KK, Akslen LA, Avril MF, Azizi E, Bakker B, Benediktsdottir KR, Bergman W, Scarra GB, Brown KM, Calista D, Chaudru V, Fargnoli MC, Cust AE, Demenais F, de Waal AC, Debniak T, Elder DE, Friedman E, Galan P, Ghiorzo P, Gillanders EM, Goldstein AM, Gruis NA, Hansson J, Helsing P, Hocevar M, Hoiom V, Hopper JL, Ingvar C, Janssen M, Jenkins MA, Kanetsky PA, Kiemeney LA, Lang J, Lathrop GM, Leachman S, Lee JE, Lubinski J, Mackie RM, Mann GJ, Martin NG, Mayordomo JI, Molven A, Mulder S, Nagore E, Novakovic S, Okamoto I, Olafsson JH, Olsson H, Pehamberger H, Peris K, Grasa MP, Planelles D, Puig S, Puig-Butille JA, Randerson-Moor J, Requena C, Rivoltini L, Rodolfo M, Santinami M, Sigurgeirsson B, Snowden H, Song F, Sulem P, Thorisdottir K, Tuominen R, Van Belle P, van der Stoep N, van Rossum MM, Wei Q, Wendt J, Zelenika D, Zhang M, Landi MT, Thorleifsson G, Bishop DT, Amos CI, Hayward NK, Stefansson K, Bishop JA, Barrett JH; GenoMEL Consortium; Q-MEGA and AMFS Investigators. A variant in FTO shows association with melanoma risk not due to BMI. Nat Genet. 2013 Apr;45(4):428-32, 432e1. doi: 10.1038/ng.2571. Epub 2013 Mar 3. PMID 23455637
- [Background] Yang XR, Rotunno M, Xiao Y, Ingvar C, Helgadottir H, Pastorino L, van Doorn R, Bennett H, Graham C, Sampson JN, Malasky M, Vogt A, Zhu B, Bianchi-Scarra G, Bruno W, Queirolo P, Fornarini G, Hansson J, Tuominen R, Burdett L, Hicks B, Hutchinson A, Jones K, Yeager M, Chanock SJ, Landi MT, Hoiom V, Olsson H, Gruis N, Ghiorzo P, Tucker MA, Goldstein AM. Multiple rare variants in high-risk pancreatic cancer-related genes may increase risk for pancreatic cancer in a subset of patients with and without germline CDKN2A mutations. Hum Genet. 2016 Nov;135(11):1241-1249. doi: 10.1007/s00439-016-1715-1. Epub 2016 Jul 23. PMID 27449771